CLINICAL TRIAL: NCT01551550
Title: Amniotic Membrane Versus Pericardium in Reducing Glaucoma Drainage Tube Exposure: A Randomized Clinical Trial
Brief Title: Shunt Tube Exposure Prevention Study
Acronym: STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Collaborators: National Eye Institute (NEI) (NIH); Bascom Palmer Eye Institute (Other); The New York Eye & Ear Infirmary (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P010-2, Version 4; R44EY019785 (NIH)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma
Keywords: Glaucoma Drainage Device, Tube Exposure, Amniotic Membrane
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants; Tutoplast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GDD & Amniotic Membrane Graft (Experimental): After GDD implantation, amniotic membrane graft (AmnioGuard™, Bio-Tissue inc, Miami, FL) is used to cover the GDD tube.
  Interventions: Procedure: GDD; Procedure: Amniotic Membrane Graft
- GDD & Pericardial Graft (Active Comparator): After GDD implantation, a pericardial graft (Tutoplast®, IOP Inc, Costa Mesa, CA) is used to cover the GDD tube.
  Interventions: Procedure: GDD; Procedure: Pericardial Graft

INTERVENTIONS:
Procedure: GDD — The surgery includes conjunctival incision, placement and securing the GDD plate in one quadrant, paracentesis and tube insertion into the anterior chamber, tube fixation to the episclera.
  Other Names: Glaucoma drainage device; Tube shunt; Shunt tube; Ahmed Valve; Baerveldt valve
Procedure: Amniotic Membrane Graft — For subjects assigned to the treatment group, Amnioguard is used to cover the shunt tube. The conjunctiva is then closed.
  Other Names: Amnioguard
  Arms: GDD & Amniotic Membrane Graft
Procedure: Pericardial Graft — For subjects assigned to the control group Tutoplast is used to cover the tube. The conjunctiva is then closed.
  Other Names: Tutoplast
  Arms: GDD & Pericardial Graft

SUMMARY:
This is a multi-site randomized clinical trial to evaluate the long-term efficacy of the thicker amniotic membrane graft (AmnioGuard™, Bio-Tissue, Inc, Miami, FL) in reducing shunt tube exposure in patients undergoing glaucoma drainage device implantation.

DETAILED DESCRIPTION:
Glaucoma drainage devices (GDDs) have been used in the treatment of high-risk refractory glaucoma. To avoid tube exposure, which may lead to serious eye infection, the implanted GDD tube must be covered by a patch graft, traditionally made of either donor sclera or pericardium. However, these patch grafts still carry a high rate of progressive thinning and erosion, a complication that the investigators speculate results from the lack of cellular infiltration from the surrounding host conjunctival stroma and poor integration of these patch grafts to the host tissue. The investigators further speculate that a thicker version of cryo-preserved amniotic membrane (AM), manufactured by Bio-Tissue, Inc.,could offer better tensile strength, be suitable for tectonic support, and have biological activities to promote cellular infiltration by the surrounding host conjunctival stroma, thus reducing progressive allogeneic patch graft thinning/erosion.

Through SBIR Phase I grant support (R43 EY19785), the investigators have evaluated the thicker AM as an alternative patch graft for covering the GDD tube during the primary implantation. The investigators further monitored the host cell interaction using anterior segment optical coherence tomography (OCT). The investigators have successfully accomplished the proposed aims of the above studies, which demonstrated the short-term stability/efficacy of AM in covering the tube in primary GDD surgery (Phase I-Aim 1) and confirmed the feasibility of using OCT to distinguish host cell infiltration into the AM after transplantation over the GDD tube (Phase I-Aim 2).

In this SBIR Phase II, the investigators propose to conduct a prospective, controlled study to compare the long-term safety and efficacy of the thicker AM (AmnioGuard™, Bio-Tissue, Inc, Miami, FL) to the pericardium (Tutoplast®, IOP Inc, Costa Mesa, CA) in securing the GDD tube and reducing tube exposure and graft thinning in patients with high risk glaucoma. The investigators will also study the risk factors that may contribute to GDD tube exposure.

Accomplishment of this Phase II study will position AM as an effective alternative to the existing patch grafts to reduce tube exposure and enhance the success of GDD implantation, while providing a better aesthetic appearance and allowing visualization of the tube in patients with high risk glaucoma. The investigators speculate that such a graft might also have other clinical applications outside of covering GDD tubes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled glaucoma undergoing GDD implantation and carry one of the following two strata of high risk factors:

  1. Primary open angle glaucoma with previous conjunctival cutting surgery including prior failed trabeculectomy.
  2. Secondary glaucoma, e.g., neovascular, uveitic, or post-traumatic glaucoma.
* Age range: 21- 80 years old.
* Both genders and all ethnic groups comparable with the local community.
* Patients able and willing to cooperate with investigational plan.
* Patients able and willing to complete postoperative follow-up.
* Patients able to understand and willing to sign a written informed consent.

Exclusion Criteria:

* Ocular infection within 14 days prior to prior to study entry.
* No light perception vision
* Previous cyclodestructive procedure.
* Children under 21 (see Inclusion of Children).
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2019-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hosam El Sheha, MD, PhD, Principal Investigator — BioTissue Holdings, Inc
Locations (4):
- United States (4):
  - Bascom Palmer Eye Institute, Miami, Florida
  - New York Eye and Ear Infirmary, New York, New York
  - Manhattan Eye, Ear, and Throat Hospital, New York, New York
  - Harkness Eye Institute/ Columbia University, New York, New York

REFERENCES:
- [Result] Anand A, Sheha H, Teng CC, Liebmann JM, Ritch R, Tello C. Use of amniotic membrane graft in glaucoma shunt surgery. Ophthalmic Surg Lasers Imaging. 2011 May-Jun;42(3):184-9. doi: 10.3928/15428877-20110426-01. PMID 21563743

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GDD & Amniotic Membrane Graft | GDD & Pericardial Graft
Started | 41 | 41
Completed | 41 | 40
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDD & Amniotic Membrane Graft | GDD & Pericardial Graft | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: yrs] | 65.4 (13.6) | 68.9 (12.3) | 67 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 19 | 12 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 10 | 28
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tube Erosion
Description: Impending conjunctival erosion can be indicated by loss of conjunctival capillaries over the tube, usually 1 to 3 mm from the corneoscleral junction. Definitive tube exposure is accompanied by conjunctival tissue loss, graft melting.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GDD & Amniotic Membrane Graft | GDD & Pericardial Graft
Number analyzed (Participants) | 41 | 40
Participants | 2 | 11

2. Secondary Outcome: Number of Participants With Glaucoma Drainage Device Failure
Description: GDD Failure, based on reoperation to control the IOP, and also include the defined by the following criteria: (1) IOP ≥21 mm Hg or not reduced by 30% below baseline on two consecutive follow-up visits after 3 months. (2) IOP ≤5 mm Hg on two consecutive follow-up visits after 3 months. (3) Additional glaucoma surgery. (4) Loss of light perception vision.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GDD & Amniotic Membrane Graft | GDD & Pericardial Graft
Number analyzed (Participants) | 41 | 40
Participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | GDD & Amniotic Membrane Graft | GDD & Pericardial Graft
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 2/41 | 3/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GDD & Amniotic Membrane Graft (N=41) | GDD & Pericardial Graft (N=41)
Corneal Edema (Eye disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No